CLINICAL TRIAL: NCT01448759
Title: Prospective Evaluation of Plasma Alcohol Concentration in Patients Receiving Paclitaxel or Docetaxel Infusion
Brief Title: Evaluation of Plasma Alcohol Concentration in Patients Receiving Paclitaxel or Docetaxel
Acronym: ALCOOTAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IC 2011-03
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Tumors
Keywords: Patients receiving docetaxel or paclitaxel. All tumors.
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood sampling — Other: Blood sampling 10mL of peripherical blood will be collected specially for the study. It's an additional blood sampling compare to the normal follow up of the patient.

SUMMARY:
The purpose of this study is to evaluate plasma alcohol concentration in patients receiving Paclitaxel or Docetaxel infusion.

DETAILED DESCRIPTION:
In this study, there is no experimental treatment, or experimental care.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy with docetaxel or paclitaxel on an every 3-week schedule.
* Patient with bitherapy are eligible only if the taxane is the first infusion.
* All type of tumor.
* Age>18 years old.
* Signed written informed consent.

Exclusion Criteria:

* Patient under 18.
* Patient with bitherapy, if docetaxel or paclitaxel is not administered first.
* Patient deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of plasma alcohol | One year
  Measure of the plasma alcohol level before and after a taxane-based therapy (docetaxel or paclitaxel)

CONTACTS AND LOCATIONS:
Overall Officials: LE TOURNEAU Christophe, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France